CLINICAL TRIAL: NCT07230028
Title: A Monocenter, Randomized, Double Blind Pilot Study Comparing Doxycycline in Combination With Hydroxychloroquine Treatment Versus Doxycycline Monotherapy in Patients With Long-Term Complaints Attributed to Lyme Borreliosis.
Brief Title: Doxycycline Boosted Therapy in Lyme Borreliosis: DoBo Study.
Acronym: DoBo
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ministerie van Volksgezondheid, Welzijn en Sport (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DoBo; 2025-523078-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-17; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Lyme Borreliosis, Nervous System
Keywords: Hydroxychloroquine
MeSH Terms: conditions — Lyme Neuroborreliosis | interventions — Hydroxychloroquine; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline in combination with Hydroxychloroquine (Experimental): Doxycycline (standard of care) in combination with Hydroxychloroquine 2 x 200 mg (two times a day one tablet).
  Interventions: Drug: Hydroxychloroquin; Drug: Doxycycline
- Doxycycline in combination with placebo (Placebo Comparator): Doxycycline (standard of care) in combination with Placebo (two times a day one tablet).
  Interventions: Drug: Placebo; Drug: Doxycycline

INTERVENTIONS:
Drug: Hydroxychloroquin — Added to the standard of care for Lyme Disease
  Other Names: Plaquenil
  Arms: Doxycycline in combination with Hydroxychloroquine
Drug: Placebo — Standard of care in combination with placebo
  Arms: Doxycycline in combination with placebo
Drug: Doxycycline — Standard of care

SUMMARY:
The goal of this clinical trial is to learn if hydroxychloroquine works to treat long-term complaints attributed to Lyme borreliosis in adults. The main questions it aims to answer are:

Does addition of hydroxychloroquine reduce physical complaints? Researchers will compare hydroxychloroquine to a placebo (a look-alike substance that contains no drug) to see if hydroxychloroquine works to treat Lyme borreliosis.

Participants will:

Take hydroxychloroquine or a placebo two times a day during 28 days. Visit the clinic 4 times in one year for checkups and tests.

DETAILED DESCRIPTION:
Rationale Assess other strategies for Lyme patients with vexing symptoms.

Objective Provide initial insights as to whether addition of hydroxychloroquine results in reduction of physical complaints and assessing safety and tolerability of hydroxychloroquine in these patients.

Main trial endpoints The primary endpoint is health-related quality of life, as measured by the global score of the 36-item Short-form General Health Survey (SF-36) at EOT (week 4).

Secondary trial endpoints Secondary endpoints are improvement on subscales of SF-36 (pain and physical function) at week 4, safety at week 4 and 12 and global physical health composite score of the 36-item Short-form General Health Survey (SF-36) at week 52. Of note, there are no biochemical or microbiological test available to assess cure.

Trial design This is a monocentre, randomized, double blind pilot study. Treatment last one month, with a follow up at week 52. In total the subject are participating for one year.

Trial population Patients with possible persisting B. burgdorferi s.l. infection or probable or possible post Lyme treatment Lyme borreliosis syndrome (PTLBS) will be recruited. Patients who will start antibiotic treatment can be included.

Interventions The intervention group will be treated with 28 days Doxycycline 2 x 100 mg (standard of care) combined with hydroxychloroquine 2 x 200 mg (two time a day one tablet). The control arm receives 28 days Doxycycline 2 x 100 mg (standard of care) combined with placebo 2 x 1 tablet.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks The combination of doxycycline en hydroxychloroquine is based on expected synergy and probably enhancement of effective therapy. Its combination has been used for years in malaria and Q-fever. Its pro- and con's are well known.

The use of doxycycline and hydroxychloroquine is not associated with increased health risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older
* Patients with probable or possible signs and symptoms attributed to Lyme borreliosis
* Patients with probable or possible post Lyme treatment Lyme borreliosis syndrome (PTLBS)
* Males or non-pregnant females (who must agree to use barrier methods of contraception during the study therapy period, women of childbearing age must have a negative urine pregnancy or serum test at baseline).

Exclusion Criteria:

* Known contra-indication for used study medication.
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life. | Week 4
  Global physical health composite score of the 36-item Short-form General Health Survey (SF-36). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. Higher scores indicating better health and lower scores indicating worse health or disability

SECONDARY OUTCOMES:
Safety of the study medication | Week 4 and week 12
  ATL (U/L), creat (μmol/L) and adverse events
Tolerability of the study medication | Week 4 and week 12
  Improvement on subscales of SF-36 questionnaire (Pain and physical function). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. higher scores indicating better health and lower scores indicating worse health or disability.
Health-related quality of life | Week 52
  Global physical health composite score of the 36-item Short-form General Health Survey (SF-36). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. Higher scores indicating better health and lower scores indicating worse health or disability

CONTACTS AND LOCATIONS:
Overall Officials: Hadewych Ter Hofstede, Dr., Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No